CLINICAL TRIAL: NCT04096313
Title: Allegro Evaluation Study for FDA Submission
Brief Title: Evaluation of the Analytical Performance of ALLEGRO™ Instrument
Status: Completed | Type: Observational
Sponsor: Nova Biomedical (Industry)
Responsible Party: Sponsor
Other Study IDs: NB19-ALL-NA-FDA
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus; Kidney Diseases; Metabolic Disease
Keywords: HbA1c, Lipids, UACR
MeSH Terms: conditions — Diabetes Mellitus; Kidney Diseases; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: HbA1c, Lipids, UACR — compare diagnostic tests to reference methods

SUMMARY:
To assess the performance of the Allegro in the hands of CLIA-Waived Point-of-Care users in at least three distinct Point-of-Care clinical settings and compare the performance characteristics to other accepted Point-of-Care methods and central laboratory reference methods.

To assess the Ease of Use of the Allegro in the hands of the intended CLIA-Waived Point-of-Care users. CLIA-Waived operators will be provided with all package insert sheets, a Quick Reference Guide poster and Instructions for Use. No training, coaching, or prompting will be provided other than clarifying the protocol.

DETAILED DESCRIPTION:
Blood and urine tests are used in the assessment of diabetes and to guide clinical management. In the traditional model of care, blood samples are taken from patients at the clinic and are sent to the laboratory for analysis and the results may not be available for a number of hours/days after the clinic visit.

A new analyser has been developed (Allegro™) which allows the tests to be undertaken at the clinic, with the results available in a few minutes. This means that patients can get immediate feedback and that the doctors/nurses can adjust treatment before the patient leaves the clinic. It is obviously important that this analyzer performs to a similar degree of accuracy to the laboratory analyses.

The aim of this research study is to assess the accuracy of the Allegro™ analyzer compared to laboratory analyses on capillary and venous whole blood samples and urine samples. Three hundred sixty (360) patients with diabetes will be invited to give a venous blood sample, finger prick capillary blood sample and urine sample. The venous blood sample, finger prick capillary blood sample and urine sample will be analysed by both the Allegro™ analyser and laboratory analyses and the results compared. The Allegro™ results will not be used in the management of the patients' diabetes.

ELIGIBILITY:
Inclusion Criteria:

* patients with ordered HbA1c, lipid profile, and UACr

Exclusion Criteria:

* pediatric

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult diabetic population
Sampling Method: Non-Probability Sample
Enrollment: 628 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Analytical verification of Allegro - HbA1c comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for HbA1c blood results in % (percentage)
Analytical verification of Allegro - Cholesterol comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for Cholesterol blood results in mg/dL
Analytical verification of Allegro - HDL comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for HDL Cholesterol blood results in mg/dL
Analytical verification of Allegro - Triglycerides comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for Triglycerides blood results in mg/dL
Analytical verification of Allegro - Urine creatinine comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for Creatinine urine results in mg/dL
Analytical verification of Allegro - Urine Albumin comparison | 10 minutes
  Allegro™, a point of care testing instrument is as effective as a reference laboratory method for Albumin urine results in g/L

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Surowitz, Principal Investigator — Health Awareness, Inc; Allison Blomer, MA, MD, Principal Investigator — Health Awareness, Inc PSL; Jeremy Bleicher, Principal Investigator — South Florida Research Organization
Locations (3):
- United States (3):
  - Health Awareness, Inc, Jupiter, Florida
  - South Florida Research Organization, Medley, Florida
  - Health Awareness, Inc PSL, Port Saint Lucie, Florida

IPD SHARING:
Plan to Share IPD: No